CLINICAL TRIAL: NCT05749536
Title: Procaterol in Elite Athletes - a PK Study
Brief Title: Pharmacokinetics of Procaterol in Elite Athletes
Acronym: Procat
Status: Completed | Type: Observational
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Vibeke Backer, professor, Bispebjerg Hospital
Other Study IDs: Procaterol
Record Dates: First submitted 2013-11-05; First posted 2023-03-01 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Asthma
Keywords: elite athletes
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — PK study
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Asthma: With positive asthma test
- Healthy: With no signs of asthma

SUMMARY:
The purpose of the study is to find blood and urine concentrations of procaterol administrated either by inhalation or by tablets in asthmatic and non-asthmatics males. We hypotheis that the concentrations of procaterol in the blood and serum is higher after tablet intake versus inhalation.

DETAILED DESCRIPTION:
Doping study

ELIGIBILITY:
Inclusion Criteria:

* Doctor diagnosed asthma for the asthmatic group
* GINA 1-3 for the asthmatic group
* Use of beta2-agonist for at least 12 months for the asthmatic group
* age 18-45
* males
* informed consent

Exclusion Criteria:

* smoker or former smoker
* airway infection to weeks prior to the study or during the study
* other chronic diseaes than asthma and allergy
* Use of beta2-agonist 6 days prior to the study
* Allergy to the study medicine

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Asthmatic and healthy volunteers
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
urine concentration of drug 0-24 h | 7 days
  In healthy subjects to investigate drug farmakokenetic
serum concentration of drug 0-24 h | 7 days
  In healthy subjects to investigate drug farmakokenetic

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke Backer, MD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Denmark